CLINICAL TRIAL: NCT01709981
Title: Anti-inflammatory Effects of Colchicine in Patients Undergoing Percutaneous Coronary Intervention: Inflammatory Marker Substudy of the Colchicine-PCI Trial
Brief Title: Anti-inflammatory Effects of Colchicine in PCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-02573
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Colchicine (Experimental): 1.2mg colchicine 1 to 2 hours prior PCI, followed by 0.6mg one hour later
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): Placebo 1-2 hours prior PCI, followed by placebo 1 hour later
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — Colchicine 1.2mg 1 to 2 hours prior PCI, followed by 0.6mg 1 hour later
  Other Names: Colcrys
  Arms: Colchicine
Drug: Placebo — Placebo 1 to 2 hours prior PCI, followed by Placebo 1 hour later
  Arms: Placebo

SUMMARY:
Peri-procedural inflammation is associated with increased rates of post-procedural myocardial infarction (MI), which occur in up to 35% of PCI patients and are themselves associated with increased risk of later MI and death. Statins suppress both inflammatory markers and MI rates during and after PCI, but ≥ 40% of PCI patients go statin-untreated, due in part to side effects such as myalgia. Moreover, because their mechanism of action relies on post-translational effects, statins must be given ≥ 12 to 24 hours prior to PCI, a time frame that is not always feasible. The investigators propose a novel alternative approach to reduce inflammation during PCI employing colchicine, an anti-inflammatory medication used frequently in gout and pericarditis. Colchicine may be particularly applicable to the PCI setting due to its rapid onset of action and excellent side-effect profile at low doses, as well as its known mechanisms of action. However, data on colchicine use in patients with coronary disease is extremely limited, and no studies to date have evaluated the use of colchicine in patients undergoing PCI. The investigators aim to characterize a potential mechanism of benefit in patients undergoing PCI by evaluating the effects of colchicine on soluble and leukocyte surface markers after PCI. The investigators also aim to determine the effects of colchicine on peri-procedural myonecrosis and MI. Accordingly, the investigators propose a prospective randomized study to characterize the effect of colchicine on inflammation and peri-procedural myocnecrosis. Patients referred for possible PCI will be randomized in a double-blinded fashion to placebo or colchicine (1.2mg 1 to 2 hours before PCI, followed by 0.6mg 1 hour later). The primary endpoint will be post-procedural interleukin-6 level. Secondary endpoints will include other relevant soluble and leukocyte-associated inflammatory markers. Sample size needed is 200 patients undergoing PCI. To adjust for a floor effect, 280 patients undergoing PCI will be needed. 400 patients will likely be needed to be enrolled to reach 280 PCIs (the remaining will have undergone a diagnostic only procedure). Of note, this is a substudy of the COLCHICINE-PCI trial (NCT 02594111)

ELIGIBILITY:
Inclusion Criteria:

* Patients must be more than 18 years of age and referred for coronary angiography

Exclusion Criteria:

* Plan for diagnostic-only coronary angiography
* On colchicine chronically
* History of intolerance to colchicine
* Glomerular filtration rate <30mL/minute or on dialysis
* Active malignancy or infection
* History of myelodysplasia
* High-dose statin load <24 hours prior to procedure
* Use of oral steroids or non-steroidal anti-inflammatory agents other than aspirin within 72 hours or 3 times the agent's half-life (whichever is longer)
* Use of strong CYP3A4/P-glycoprotein inhibitors (specifically ritonavir, ketoconazole, clarithromycin, cyclosporine, diltiazem and verapamil)
* Unable to consent
* Participating in a competing study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2013-05-30 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Binita Shah, MD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - Manhattan VA Hospital, New York, New York
  - Bellevue Hospital Center, New York, New York
  - New York Langone Medical Center, New York, New York

REFERENCES:
- [Derived] Shah B, Pillinger M, Zhong H, Cronstein B, Xia Y, Lorin JD, Smilowitz NR, Feit F, Ratnapala N, Keller NM, Katz SD. Effects of Acute Colchicine Administration Prior to Percutaneous Coronary Intervention: COLCHICINE-PCI Randomized Trial. Circ Cardiovasc Interv. 2020 Apr;13(4):e008717. doi: 10.1161/CIRCINTERVENTIONS.119.008717. Epub 2020 Apr 16. PMID 32295417

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Colchicine | Placebo
Started | 141 | 139
Completed | 141 | 139
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Colchicine: Colchicine
- Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Colchicine | Placebo | Total
Number analyzed (Participants) | 141 | 139 | 280
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.31 (9.29) | 65.15 (10.38) | 64.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 130 | 127 | 257
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 30 | 64
  Not Hispanic or Latino | 107 | 109 | 216
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 11 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 25 | 57
  White | 105 | 102 | 207
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 141 | 139 | 280

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Post-procedural IL-6 Concentration From Baseline to 30 Min -1 hr After PCI
Time Frame: 30 minutes to 1 hour after PCI
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 140 | 138
% change | 0 [-161 to 241] | 20 [-99 to 282]
Statistical Analysis 1: Comparison: Colchicine vs Placebo; Test type: Equivalence — Mann-Whitney; p = 0.31, Wilcoxon (Mann-Whitney); 2-sided

2. Secondary Outcome: Percent Change in Post-procedural IL-6 Concentration From Baseline to 22-24 hr After PCI
Time Frame: baseline to 22-24 hr after PCI
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 120 | 122
% change | 76 [-6 to 898] | 338 [27 to 1264]

3. Secondary Outcome: Percent Change in Post-procedural hsCRP Concentration From Baseline to 22-24 hr After PCI
Time Frame: baseline to 22-24 hr after PCI
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 123 | 124
% change | 11 [-14 to 80] | 66 [1 to 172]

4. Secondary Outcome: Percent Change in Post-procedural IL-1B Concentration From Baseline to 30 Min -1 hr After PCI
Time Frame: 30 minutes to 1 hour after PCI
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 140 | 138
% change | 0 [-2 to 9] | 0 [-5 to 7]

5. Secondary Outcome: Percent Change in Post-procedural IL-1B Concentration From Baseline to 30 Min -1 hr After PCI
Time Frame: baseline to 22-24 hr after PCI
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 120 | 122
% change | 0 [0 to 8] | 0 [-9 to 6]

ADVERSE EVENTS:
Time Frame: 30 days, 6 months, and yearly for 5 years
Arm/Group | Colchicine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/139
Serious Adverse Events (participants affected / at risk) | 2/141 | 6/139
Other Adverse Events (participants affected / at risk) | 0/141 | 0/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colchicine (N=141) | Placebo (N=139)
Chest pain (Cardiac disorders) | 1 (1) | 1 (1)
Ischemic stroke (Vascular disorders) | 1 (1) | 0 (0)
Fever (Immune system disorders) | 0 (0) | 1 (1)
Hemodynamic instabiity (General disorders) | 0 (0) | 2 (2)
Elevated creatinine (Renal and urinary disorders) | 0 (0) | 1 (1)
Bleeding (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT01709981/Prot_003.pdf
  • Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT01709981/SAP_002.pdf